CLINICAL TRIAL: NCT06405087
Title: A Phase 3b Extension Study to Evaluate the Long-term Safety of Vedolizumab Subcutaneous in Pediatric Subjects With Ulcerative Colitis or Crohn's Disease
Brief Title: A Long-Term Extension Study of Vedolizumab in Children and Teenagers With Ulcerative Colitis (UC) or Crohn's Disease (CD)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VedolizumabSC-3004; 2023-508804-39-00 (EU CTIS Number: EU CT Number); jRCT2031250519 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis; Crohn's Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Cohort: Vedolizumab 108 mg PFS+AI (Experimental): Vedolizumab 108 mg, PFS+AI, subcutaneously, once every two weeks (Q2W) to the participants weighing greater than or equal to (>=) 30 kg and once every four weeks (Q4W) to the participants weighing >=10 to less than (<) 30 from Day 1 up to Week 120, until participant withdraws from the study, or until vedolizumab SC is commercially available for pediatric indication in the participant's country or other drug access programs become available, or the sponsor decides to close the study, whichever occurs first.
  Interventions: Drug: Vedolizumab SC
- Treatment Cohort: Vedolizumab 108 mg PFS+NSD (Experimental): Vedolizumab 108 mg, PFS+NSD, subcutaneously, Q2W to the participants weighing >=30 kg and Q4W to the participants weighing >=10 to <30 from Day 1 up to Week 120, until participant withdraws from the study, or until vedolizumab SC is commercially available for pediatric indication in the participant's country or other drug access programs become available, or the sponsor decides to close the study, whichever occurs first.
  Interventions: Drug: Vedolizumab SC
- Observational Cohort: Early Terminated Participants From Parent Study (Other): Participants who receive any dose of vedolizumab SC during the parent study VedolizumabSC-3003 (NCT06100289) and are not eligible for the treatment cohort of this extension study (that is, participants who early terminated from parent study VedolizumabSC-3003 [NCT06100289] or did not achieve clinical response in the parent study or who received corticosteroids in the last 4 weeks of the parent study) will only be observed in the observational cohort of this study and will not receive any dose of the vedolizumab SC in this cohort.
  Interventions: Other: No Intervention

INTERVENTIONS:
Drug: Vedolizumab SC — Vedolizumab subcutaneous injection.
  Other Names: MLN0002
  Arms: Treatment Cohort: Vedolizumab 108 mg PFS+AI; Treatment Cohort: Vedolizumab 108 mg PFS+NSD
Other: No Intervention — As this is an observational cohort, no intervention will be administered.
  Arms: Observational Cohort: Early Terminated Participants From Parent Study

SUMMARY:
The main aim of this study is to learn about medical problems (adverse events) if vedolizumab subcutaneously (SC) is given to a child or teenager with UC or CD for a long time. Other aims are to understand if the long time use of vedolizumab SC has an impact on the time period until hospital visits because of bowel swelling (inflammation) are needed and has an impact on the quality of life of children and teenagers who received vedolizumab SC.

In this study, participants who responded well to the treatment with vedolizumab SC in the parent study (VedolizumabSC-3003 [NCT06100289]) will continue to be treated with vedolizumab SC. Participants who did not respond well to the treatment with vedolizumab SC in the parent study or who received corticosteroids in the last 4 weeks of the parent study will not receive vedolizumab SC in this study but will be followed for up to 2 years after the last treatment with vedolizumab SC in the parent study.

During the study, participants will visit their study clinic several times.

DETAILED DESCRIPTION:
The drug being tested in this study is Vedolizumab SC. Vedolizumab SC is being tested to treat pediatric participants with moderate to severe active UC or CD. This study will look at the long-term safety profile in pediatric participants who take vedolizumab SC.

The study will enroll approximately 70 participants. This extension study consists of a treatment cohort and an observational cohort. Participants will continue receiving the same dose and frequency of vedolizumab SC that was received at the last dose of the parent study VedolizumabSC-3003 (NCT06100289).

For the Treatment cohort participants will be randomized (1:1) to receive vedolizumab in either a prefilled syringe (PFS) as part of an autoinjector pen (PFS+AI) or a PFS with a needle safety device (PFS+NSD):

* Treatment Cohort: Vedolizumab 108 milligram (mg) PFS+AI
* Treatment Cohort: Vedolizumab 108 mg PFS+NSD

This multi-center trial will be conducted globally. The overall time to participate in this study is up to 2 years from the first dose in the study. Participants in the treatment cohort will have a follow-up safety visit of 18 weeks after their last dose of study drug. Participants who will not be eligible for the treatment cohort will be enrolled in the observational cohort and will be followed for approximately 2 years after the last dose of vedolizumab SC received during Study VedolizumabSC-3003 (NCT06100289).

ELIGIBILITY:
Inclusion Criteria for Treatment Cohort 1. Has completed Week 34 of Study VedolizumabSC-3003 (NCT06100289) and achieved clinical response at Week 34 and was corticosteroid-free for at least the last 4 weeks (Week 30 to Week 34). Clinical response for participants with UC is defined as a reduction of partial Mayo score of >=2 points and >= 25 percentage (%) from baseline (from VedolizumabSC-3003 [NCT06100289]), including a >=1-point decrease in the Mayo stool frequency subscore and a >=1-point reduction in the rectal bleeding subscore or absolute rectal bleeding subscore of less than or equal to (<=) 1 point. Clinical response for participants with CD is defined as a pediatric Crohn's disease activity index (PCDAI) <=30 with a reduction in the PCDAI of >=15 points from baseline (from VedolizumabSC-3003 [NCT06100289]).

Inclusion Criteria for Observational Cohort

1. Has received at least 1 dose of vedolizumab during Study VedolizumabSC-3003 (NCT06100289) and early terminated OR completed the Week 34 clinic visit of Study VedolizumabSC-3003 (NCT06100289) but was not eligible to enroll in the treatment cohort of this study.

Exclusion Criteria for Treatment Cohort

1. Has hypersensitivity or allergies to vedolizumab or any of its excipients.
2. The participant currently requires major surgical intervention for UC or CD (example, bowel resection), or is anticipated to require major surgical intervention for UC or CD during the study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2032-01-26 (Estimated); Study Completion 2032-01-26 (Estimated)

PRIMARY OUTCOMES:
Treatment Cohort: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | First dose of the study drug until 18 weeks of follow-up after last dose (up to Week 138)
  An Adverse event (AE) is defined as any untoward medical occurrence in clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory value), symptom, or disease temporally associated with use of drug whether or not it is considered related to drug. SAE is defined as any untoward medical occurrence that at any dose: results in death, is life threatening.
Treatment Cohort: Number of Participants With Adverse Events of Special Interests (AESIs) | First dose of the study drug until 18 weeks of follow-up after last dose (up to Week 138)
  AESI is defined as infections, including opportunistic infection, such as progressive multifocal leukoencephalopathy (PML), liver injury, malignancies, injection-related reactions or systemic reactions including anaphylaxis and hypersensitivity reactions.
Observational Cohort: Number of Participants With Prespecified Safety Events | Up to Week 86
  Prespecified safety events will include serious infections, malignancies, PML, concerns about growth and pubertal development, and bowel surgery.

SECONDARY OUTCOMES:
Treatment Cohort: Time to Major Inflammatory Bowel Disease (IBD)-related Events | Up to Week 120
  Time to major IBD related events is defined as time to first occurrence of any among the 3 IBD related events such as: hospitalizations, surgeries, and procedures.
Treatment Cohort: Change from Baseline in IMPACT-III Scores | Baseline, every 24 weeks in this study (up to Week 120)
  IMPACT-III questionnaire will be administered to participants aged 9 to 17 years. The IMPACT-III questionnaire is a self-reported measure with 35 closed questions encompassing 6 domains: Bowel Symptoms (7 items), Systemic Symptoms (3 items), Social Functioning (12 items), Body Image (3 items), Treatment/Interventions (3 items), and Emotional Functioning (7 items). The IMPACT-III uses a 5-point Likert subscale score ranging from 1 to 5 for all answers. The outcome total score ranges from 35 to 175, with higher scores suggesting better quality of life. Baseline refers to the Baseline of study VedolizumabSC-3003 (NCT06100289).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Juntendo University Hospital, Bunkyo-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/e43dc491502443a5??page=1&idFilter=VedolizumabSC-3004